CLINICAL TRIAL: NCT02950467
Title: Psilocybin-assisted Group Therapy for Demoralization in Long-term AIDS Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joshua Woolley (Other)
Collaborators: Heffter Research Institute (Other); RiverStyx Foundation (Other); Usona Institute (Other); Stupski Foundation (Other)
Responsible Party: Sponsor-Investigator, Joshua Woolley, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-17825
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Distress; Depression; Grief
Keywords: HIV/AIDS; Demoralization; Psilocybin; Group therapy
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group therapy plus psilocybin (Experimental): Modified brief Supportive-Expressive Group Therapy will be administered as ten twice-weekly sessions. Oral psilocybin will be administered once in a clinical setting.
  Interventions: Drug: Psilocybin; Behavioral: Modified brief Supportive Expressive Group Therapy

INTERVENTIONS:
Drug: Psilocybin — One individual oral psilocybin treatment session
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine; Indocybin
Behavioral: Modified brief Supportive Expressive Group Therapy — Ten sessions of twice-weekly manualized group therapy

SUMMARY:
The purpose of this study is to determine whether psilocybin-assisted group psychotherapy is a safe and feasible treatment for demoralization in long-term AIDS survivors (LTAS).

DETAILED DESCRIPTION:
This study is an open-label mixed-methods pilot study of an individual oral psilocybin drug session combined with ten sessions of an evidence-based, manualized brief group psychotherapy for existential distress in palliative care patients.

ELIGIBILITY:
Inclusion Criterion:

* Older individuals who are long-term AIDS survivors and suffer from moderate-to-severe demoralization.

Exclusion Criteria:

* A physical, neurological or cognitive condition that makes participating in the study unsafe or unfeasible.
* Regular psychotropic medication use.
* Personal or family history of serious mental illness.
* Severe depression requiring immediate standard-of-care treatment.
* Exclusion by the clinical judgment of the study investigators.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD,PhD, Principal Investigator — University of California, San Francisco; Brian Anderson, MD,MSc, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson BT, Danforth A, Daroff PR, Stauffer C, Ekman E, Agin-Liebes G, Trope A, Boden MT, Dilley PJ, Mitchell J, Woolley J. Psilocybin-assisted group therapy for demoralized older long-term AIDS survivor men: An open-label safety and feasibility pilot study. EClinicalMedicine. 2020 Sep 24;27:100538. doi: 10.1016/j.eclinm.2020.100538. eCollection 2020 Oct. PMID 33150319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community 17 July 2017 to 24 August 2018 in the San Francisco Bay Area.
Pre-assignment Details: 91 study candidates were screened over the phone, of which 37 were eligible for in-person enrollment evaluations, of which 30 attended an in-person enrollment evaluation and were consented to the study. 18 candidates were found to be eligible for the study, all of whom enrolled in the trial and initiated treatment.
Period: Open-label Treatment
Arm/Group | Group Therapy Plus Psilocybin
Started | 18
Completed | 18 (1 participant completed study period but missed some visits due to an adverse event (AE).)
Not Completed | 0
Period: 3-month Follow-up
Arm/Group | Group Therapy Plus Psilocybin
Started | 18
Completed | 18 (All participants completed the safety follow-up assessment, but not all completed outcomes measures.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Year of HIV/AIDS/GRID Diagnosis [Mean (Standard Deviation); unit: years] — HIV = Human immunodeficiency virus; AIDS = Acquired immunodeficiency syndrome; GRID = Gay-related immunodeficiency
  years | 1988 (4.8)
Palliative Performance Scale v2.0 [Mean (Standard Deviation); unit: units on a scale] — This clinician-rated scale reports a total score ranging from 0% (Death) to 100% (Full ambulation, normal activity and work, full self-care, etc). Higher scores indicate better performance.
  units on a scale | 92.8 (11.3)
Civil status [Count of Participants; unit: Participants]
  Single | 8
  Married/Partnered | 8
  Divorced/Separated | 2
Education [Count of Participants; unit: Participants]
  Less than college | 5
  College or more | 13
Annual income [Count of Participants; unit: Participants]
  <$50,000 | 10
  ≥$50,000 | 8
Patients meeting current SCID-5/SCID-5-PD diagnosis [Number; unit: participants] — These diagnostic categories are not mutually exclusive. Patients may meet criteria for more than one diagnosis at one time.
  SCID = Structured Clinical Interview for DSM-5 SCID-PD = Structured Clinical Interview for DSM-5 - Personality Disorders DSM-5 = Diagnostic and Statistical Manual of Mental Disorders
  participants
    Generalized anxiety disorder | 7
    Major depressive disorder | 5
    Panic disorder | 3
    Borderline personality disorder | 3
    No SCID-5/SCID-5-PD diagnosis (of those assessed) | 9
PTSD Checklist-5 (PCL-5) >33/80 [Count of Participants; unit: Participants] — PCL-5 is a self-report checklist used to screen for PTSD symptoms. A score >33/80 indicates a possible diagnosis of current PTSD. Higher scores indicated worse PTSD severity.
  Participants | 3
Lifetime: People close to you who have died [Median (Inter-Quartile Range); unit: people] | 17.5 [7.25 to 30]
Lifetime: Times used a classic psychedelic [Median (Inter-Quartile Range); unit: instances] | 5 [3 to 23]
Years since last used a classic psychedelic [Median (Inter-Quartile Range); unit: years] | 20 [1 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-related Adverse Events as Assessed by NIH Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0
Description: Full details of adverse event data are in the Adverse Events module of this ClinicalTrials.gov entry.
  Adverse events were assessed at every study visit by patient interview. During medication visits, adverse events were also assess by vitals sign monitoring, patient self-report, and adverse events observed by clinicians.
Time Frame: Enrollment to 3-month follow up, about 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
Participants | 18

2. Primary Outcome: Subject Recruitment and Retention
Description: Two therapy groups of at least 4 subjects each will complete the study
Time Frame: Duration of study, about 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
Participants
  Enrolled | 18
  Completed Safety Assessment at End-of-treatment | 18
  Completed Safety Assessment at 3-month follow-up | 18

3. Secondary Outcome: Change From Baseline in Demoralization Scale-II at End-of-treatment
Description: Demoralization self-report measure. Minimum = 0. Maximum = 32. Higher scores means a worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -6.67 (6.5)

4. Secondary Outcome: Change From Baseline in Demoralization Scale-II at 3-month Follow-up
Description: Demoralization self-report measure. Minimum = 0. Maximum = 32. Higher scores mean a worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: Intent-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -5.78 (6.01)

5. Secondary Outcome: Change From Baseline in Inventory of Complicated Grief-Revised at End-of-treatment
Description: Complicated Grief self-report measure. Minimum = 0, Maximum = 76. Higher scores mean worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -6.22 (6.74)

6. Secondary Outcome: Change From Baseline in Inventory of Complicated Grief at 3-month Follow-up
Description: Complicated Grief self-report measure. Minimum = 0, Maximum = 76. Higher scores mean worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -7.06 (7.61)

7. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale-Revised at End-of-treatment
Description: Depression self-report measure. Minimum = 0. Maximum = 60. Higher scores mean a worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -8.94 (14.73)

8. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale-Revised at 3-month Follow-up
Description: Depression self-report measure. Minimum = 0. Maximum = 60. Higher scores mean a worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -8.89 (12.02)

9. Secondary Outcome: Change in Average Score on Subscales of Group Questionnaire Pre-drug vs Post-drug
Description: The Group Questionnaire is a self-report measure with three sub-scales that measure Positive Bonding, Positive Working and Negative Relationship dimensions of the relationships at 3 levels: between group members, between group members and group therapists, and between group members and the group as a whole. Each subscale score is calculated by summation of the ratings across all three levels for each subscale. Positive Bonding scores range from 13 to 91 with higher scores indicating a better outcome. Positive Working scores range 8 to 56 with higher scores indicating a better outcome. Negative Relationship scores range 9 to 63 with higher scores indicating worse outcomes.
Time Frame: Mean scores averaged over 2 weeks pre-medication compared to 3 weeks post-medication.
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
score on a scale
  Positive Bonding (Overall) | 2.61 (4.77)
  Positive Working (Overall) | 1.87 (7.31)
  Negative Relationship (Overall) | -0.69 (2.70)

10. Other Pre Specified Outcome: Change From Baseline in PTSD Checklist 5 at End-of-treatment
Description: PTSD self-report measure. Minimum = 0. Maximum = 80. Higher scores mean a worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -9 (11.47)

11. Other Pre Specified Outcome: Change From Baseline in PTSD Checklist 5 at 3-month Follow-up
Description: PTSD self-report measure. Minimum = 0. Maximum = 80. Higher scores mean a worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -7.11 (13.81)

12. Other Pre Specified Outcome: Change From Baseline in State-Trait Anxiety Inventory (State) at End-of-treatment
Description: State anxiety self-report measure. Minimum = 0. Maximum = 80. Higher scores mean a worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -5.56 (9.04)

13. Other Pre Specified Outcome: Change From Baseline in State-Trait Anxiety Inventory (State) at 3-month Follow-up
Description: State anxiety self-report measure. Minimum = 0. Maximum = 80. Higher scores mean a worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | 1.06 (13.23)

14. Other Pre Specified Outcome: Change From Baseline in State-Trait Anxiety Inventory (Trait) at End-of-treatment
Description: Trait anxiety self-report measure. Minimum = 0. Maximum = 80. Higher scores mean a worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -6.06 (5.5)

15. Other Pre Specified Outcome: Change From Baseline in State-Trait Anxiety Inventory (Trait) at 3-month Follow-up
Description: Trait anxiety self-report measure. Minimum = 0. Maximum = 80. Higher scores mean a worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -3.39 (10.55)

16. Other Pre Specified Outcome: Change From Baseline in HIV and Abuse Related Shame Inventory at End-of-treatment
Description: HIV-related shame self-report measure. Minimum = 0. Maximum = 52. Higher scores mean a worse outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -5.83 (5.23)

17. Other Pre Specified Outcome: Change From Baseline in HIV and Abuse Related Shame Inventory at 3-month Follow-up
Description: HIV-related shame self-report measure. Minimum = 0. Maximum = 52. Higher scores mean a worse outcome.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat (data capture error for 6 participants)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 12
units on a scale | -4.25 (4.47)

18. Other Pre Specified Outcome: Change From Baseline in Experiences in Closer Relationships-M16 (Anxiety) at End-of-treatment
Description: Self-report measure of attachment anxiety. Minimum = 8. Maximum = 56. Higher scores mean worse outcomes.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -0.78 (8.86)

19. Other Pre Specified Outcome: Change From Baseline in Experiences in Closer Relationships-M16 (Anxiety) at 3-month Follow-up
Description: Self-report measure of attachment anxiety. Minimum = 8. Maximum = 56. Higher scores mean worse outcomes.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -3.33 (7.66)

20. Other Pre Specified Outcome: Change From Baseline in Experiences in Closer Relationships-M16 (Avoidance) at End-of-treatment
Description: Self-report measure of attachment avoidance. Minimum = 8. Maximum = 56. Higher scores mean worse outcomes.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -2.72 (6.85)

21. Other Pre Specified Outcome: Change From Baseline in Experiences in Closer Relationships-M16 (Avoidance) at 3-month Follow-up
Description: Self-report measure of attachment avoidance. Minimum = 8. Maximum = 56. Higher scores mean worse outcomes.
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | -0.06 (6.3)

22. Other Pre Specified Outcome: Change From Baseline in McGill Quality of Life Questionnaired-Revised (Overall) at End-of-treatment
Description: Self-report quality of life measure. Only item A) Overall quality of life. Minimum = 0 (Very bad). Maximum = 10 (Excellent). Higher scores mean better outcomes.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | 2.0 (1.91)

23. Other Pre Specified Outcome: Change From Baseline in McGill Quality of Life Questionnaire-Revised (Overall) at 3-month Follow-up
Description: as for outcome 22
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 18
units on a scale | 0.94 (2.44)

24. Other Pre Specified Outcome: Change From Baseline in Antiretroviral Medication Adherence Scale at End-of-treatment
Description: Self-report last-month antiviral medication adherence. Minimum = 0%. Maximum = 100%. Higher scores mean a better outcome.
Time Frame: Baseline and end-of-treatment (7 weeks duration)
Population: intent-to-treat (one participant did not use antiretrovirals)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 17
units on a scale | -0.71 (4.0)

25. Other Pre Specified Outcome: Change From Baseline in Antiretroviral Medication Adherence Scale at 3-month Follow-up
Description: as for outcome 24
Time Frame: Baseline and 3-month follow-up
Population: intent-to-treat (one participant did not use antiretrovirals)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Therapy Plus Psilocybin
Number analyzed (Participants) | 17
units on a scale | -0.94 (2.38)

ADVERSE EVENTS:
Time Frame: From Baseline to 3-month follow-up (5-months post-Baseline)
Arm/Group | Group Therapy Plus Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Therapy Plus Psilocybin (N=18)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stimulant-induced psychosis (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Therapy Plus Psilocybin (N=18)
Hypertension (severe, asymptomatic) (Vascular disorders) | 4 (4)
Hypertension (moderate) (Vascular disorders) | 8 (8)
Anxiety / Anxiety Exacerbation (Psychiatric disorders) | 8 — (moderate-severe)
Nausea (Gastrointestinal disorders) | 6
Headache (Nervous system disorders) | 5
Paranoia / Ideas of Reference (Psychiatric disorders) | 4
Motor agitation / Restlessness (Nervous system disorders) | 4
Unsteady gait / Ataxia (Nervous system disorders) | 4
Tachycardia (Cardiac disorders) | 2
Thought disorder (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Visual changes (complaint) (Nervous system disorders) | 1
Headache (post-medication visit) (Nervous system disorders) | 8
Fatigue (post-medication visit) (General disorders) | 2
Insomnia (post-medication visit) (Psychiatric disorders) | 2
Anxiety exacerbation (post-medication visit) (Psychiatric disorders) | 1 — with methamphetamine lapse
Post-traumatic stress flashback (post-medication visit) (Psychiatric disorders) | 1 — with tinnitus, nausea, panic and insomnia
Nausea (post-medication visit) (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Final protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT02950467/Prot_SAP_000.pdf
  • Informed Consent Form: Final ICF (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT02950467/ICF_001.pdf
  • Informed Consent Form: ICF for Cohorts 2 and 3 (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT02950467/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan: Pre-modifications related to enrollment exceptions (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT02950467/Prot_SAP_003.pdf